CLINICAL TRIAL: NCT01141335
Title: Lichtenstein's Repair of Inguinal Hernia With Polypropylene Mesh Versus Infinit® PTFE Mesh, a Prospective Randomized, Double-blind, Controlled Trial
Brief Title: Polypropylene Mesh Versus Polytetrafluoroethylene (PTFE) Mesh in Inguinal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS-002
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Physical Function; Pain; Hernia; Wound Infection; Postoperative Complication; Recurrence
Keywords: shrinkage; postoperative pain and discomfort
MeSH Terms: conditions — Pain; Hernia; Wound Infection; Postoperative Complications; Recurrence; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTFE mesh (Experimental): A Lichtenstein tension-free hernioplasty is performed using PTFE mesh
  Interventions: Device: Infinit® PTFE mesh (WL Gore)
- polypropylene mesh (Active Comparator): A Lichtenstein tension-free hernioplasty is performed using polypropylene mesh
  Interventions: Device: polypropylene mesh

INTERVENTIONS:
Device: polypropylene mesh — A Lichtenstein tension-free hernioplasty is performed using a polypropylene mesh will be fixed by sutures in Polypropylene 2/0.
  Arms: polypropylene mesh
Device: Infinit® PTFE mesh (WL Gore) — A Lichtenstein tension-free hernioplasty is performed using a PTFE mesh will be fixed by sutures in PTFE 2/0.
  Arms: PTFE mesh

SUMMARY:
To evaluate the safety and efficacy of the Lichtenstein's hernioplasty using Infinit® PTFE Mesh, and to compare it with the traditional Lichtenstein procedure performed with polypropylene mesh.

ELIGIBILITY:
Inclusion Criteria:

* >18 <65 years of age
* Diagnosis of Unilateral inguinal hernia
* Able to provide written consent
* BMI < 35
* ASA I-II patients
* Non-complicated primary inguinal hernia performed in non-emergency setting and repaired with a Lichtenstein's hernioplasty
* Informed consent

Exclusion Criteria:

* Recurrent hernias
* Incarcerated hernia
* BMI > 35
* ASA III-IV patients
* Any condition preventing a correct evaluation of pain (non-cooperative patient, blind patient, drug addicted)
* Hypersensitivity to any drug in study
* Patients with an intra-operative findings of different pathology will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
post-hernioplasty acute pain | 24 hours
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups

SECONDARY OUTCOMES:
physical function | 24 hours
  to measure the physical function score from the SF-36 questionnaire
postoperative acute discomfort | 24 hours
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
wound infection | 7 days
  to rate the wound infection risk.
postoperative complication | from 24 hours to 5 years
  to monitor any other postoperative complication observed in the immediate, mid-term and long-term postoperative period.
recurrence | from 1 months to 5 years
  to measure the recurrence
mesh shrinkage | 14 days
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
post-hernioplasty acute pain | 72 hours
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty acute pain | 7 days
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty acute pain | 14 days
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 1 months
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 3 months
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 6 months
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 1 year
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 2 years
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 3 years
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 4 years
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
post-hernioplasty chronic pain | 5 years
  to measure the degree of post-hernioplasty acute and chronic pain with visual analogue scale (VAS), and parenteral/oral analgesic consumption in the two groups
physical function | 72 hours
  to measure the physical function score from the SF-36 questionnaire
physical function | 7 days
  to measure the physical function score from the SF-36 questionnaire
physical function | 14 days
  to measure the physical function score from the SF-36 questionnaire
physical function | 1 months
  to measure the physical function score from the SF-36 questionnaire
physical function | 3 months
  to measure the physical function score from the SF-36 questionnaire
physical function | 6 months
  to measure the physical function score from the SF-36 questionnaire
physical function | 1 year
  to measure the physical function score from the SF-36 questionnaire
physical function | 2 years
  to measure the physical function score from the SF-36 questionnaire
physical function | 3 years
  to measure the physical function score from the SF-36 questionnaire
physical function | 4 years
  to measure the physical function score from the SF-36 questionnaire
physical function | 5 years
  to measure the physical function score from the SF-36 questionnaire
postoperative acute discomfort | 72 hours
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative acute discomfort | 14 days
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 1 months
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 3 months
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 6 months
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 1 year
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 2 years
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 3 years
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 4 years
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative chronic discomfort | 5 years
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
postoperative acute and chronic discomfort | 7 days
  to measure the degree of postoperative acute and chronic discomfort with visual analogue scale (VAS).
wound infection | 14 days
  to rate the wound infection risk.
wound infection | 1 months
  to rate the wound infection risk.
wound infection | 3 months
  to rate the wound infection risk.
wound infection | 6 months
  to rate the wound infection risk.
wound infection | 1 year
  to rate the wound infection risk.
wound infection | 2 years
  to rate the wound infection risk.
wound infection | 3 years
  to rate the wound infection risk.
wound infection | 4 years
  to rate the wound infection risk.
wound infection | 5 years
  to rate the wound infection risk.
mesh shrinkage | 1 months
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 3 months
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 6 months
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 1 years
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 2 years
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 3 years
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 4 years
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound
mesh shrinkage | 5 years
  to measure the effectiveness shrinkage of the two different mesh using Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Masoni, Dr., Study Chair — Azienda Ospedaliera Sant'Andrea, Rome, Italy; Francesco Saverio Mari, Dr., Principal Investigator — Azienda Ospedaliera Sant'Andrea, Rome, Italy; Antonio Brescia, Prof., Study Director — Azienda Ospedaliera Sant'Andrea, Rome, Italy; Giuseppe R Nigri, Dr., Principal Investigator — Azienda Ospedaliera Sant'Andrea, Rome, Italy; Francesco Favi, Dr, Principal Investigator — Azienda Ospedaliera Sant'Andrea, Rome, Italy; Andrea Milillo, Dr., Principal Investigator — Azienda Ospedaliera Sant'Andrea, Rome, Italy
Locations (1):
- UO Oneday-day Surgery, Azienda Ospedaliera Sant'Andrea, Rome, Italy, Italy